CLINICAL TRIAL: NCT04430881
Title: The SMS Study, a National Study on Prevalence of Unexplained Splenomegaly Etiologies
Brief Title: A National Study in Patients With Unexplained Splenomegaly
Acronym: SMS
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: DIREGL07298
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Gaucher Disease; Splenomegaly
MeSH Terms: conditions — Gaucher Disease; Splenomegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — max 1000 characters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary Objective:

To estimate the prevalence of Gaucher disease and of other etiologies, in patients of 15 years old or more presenting with unexplained splenomegaly after exclusion of first intention-diagnoses (e.g. portal hypertension, diagnosis or suspicion of haematological malignancy, haemolytic anemia) based on basic physical and biological exams (e.g. full blood count, liver enzymes, reticulocytes)

Secondary Objective:

To describe the exams and tests conducted for diagnosis purpose and the more frequent associations

DETAILED DESCRIPTION:
Study duration per participant is between 1 and 12 months

ELIGIBILITY:
Inclusion criteria:

* Participants referred for the first time for splenomegaly exploration defined as :

  * Either a palpable mass on left upper abdominal quadrant, further confirmed by a ≥ 13 cm craniocaudal length on abdominal Imaging
  * Or a non palpable splenomegaly discovered on abdominal imaging and with a craniocaudal length ≥ 13 cm
* Participants with splenomegaly (as defined above) of unknown origin

Exclusion criteria:

* Participants with obvious diagnostics based on clinical exam, patient's interview and the previous initial routine biological tests :

  * Diagnosis of portal hypertension
  * Diagnosis of hemolytic anemia
  * Diagnosis of hematological malignancy
  * Known diagnosis of Gaucher Disease

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants of 15 years old or more presenting with unexplained splenomegaly after exclusion of first intention-diagnoses (e.g. portal hypertension, diagnosis or suspicion of haematological malignancy, haemolytic anemia) based on basic physical and biological exams
Sampling Method: Probability Sample
Enrollment: 506 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Percentage of patients diagnosed with Gaucher disease in the included population of patients with unexplained splenomegaly | between 1 and 12 months
  The diagnosis of Gaucher Disease is based on a value of beta-glucosidase enzyme activity

SECONDARY OUTCOMES:
Percentage of patients with other than Gaucher disease-etiologies in the included population | between 1 and 12 months
  These will be any etiology among all the diseases that can be considered in the differential diagnosis of unexplained splenomegaly, e.g.: infection, haematological, congestive, inflammatory, neoplastic, infiltrative, benign tumors, immune, iron deficiencies and other miscellaneous rare causes
Number of participants by type of exams and tests conducted for diagnosis purpose | between 1 and 12 months
  Relevant exams and tests performed, in each site, for the participant diagnosis other than Gaucher disease will be reported , this may include dried blood spot, medullary biopsy, imaging exploration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site France, France, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Denis G, Terriou L, Sene T, Costello R, Michaud M, Lagadec A, Bauduer F, Sanhes L, Rose C, Urbanski G, Berger MG. SplenoMegaly study (SMS): exploring the etiologies for "unexplained" splenomegalies in the real world. Orphanet J Rare Dis. 2025 Jun 6;20(1):285. doi: 10.1186/s13023-025-03768-3. PMID 40481534